CLINICAL TRIAL: NCT01291381
Title: Regulatory T Cells in the Response to SIT in Allergic Rhinitis.
Brief Title: Distinct Response of CD4+CD25+Foxp3+ and IL-10-secreting Type I T Regulatory Cells to Cluster Specific Immunotherapy in Allergic Rhinitis Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Professor Luo Zhang, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-BIO-01; 81025007 (Other Grant/Funding Number: the National Science Fund)
Record Dates: First submitted 2011-01-25; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2009-01

CONDITIONS: Allergic Rhinitis; Effects of Immunotherapy
Keywords: allergic rhinitis; peripheral tolerance; regulatory T cells; specific immunotherapy; Tr1 cells
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Antigens, Dermatophagoides; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dermatophagoides pteronyssinus extract (Active Comparator): Children undergoing subcutaneous immunotherapy were given Dermatophagoides pteronyssinus extract (Alutard SQ, ALK-Abello, Hørsholm, Denmark) according to a cluster protocol
  Interventions: Drug: Dermatophagoides pteronyssinus
- Pharmacotherapy (Active Comparator): Persistent rhinitis was managed with pharmacotherapy including intranasal steroids and oral antihistamines. Intranasal steroids were kept at the same dose during the study and antihistamines were used as required.
  Interventions: Drug: Pharmacotherapy

INTERVENTIONS:
Drug: Dermatophagoides pteronyssinus — Children undergoing subcutaneous immunotherapy were given Dermatophagoides pteronyssinus extract (Alutard SQ, ALK-Abello, Hørsholm, Denmark) according to a cluster protocol
  Arms: Dermatophagoides pteronyssinus extract
Drug: Pharmacotherapy — For patients randomized to non-SIT group, persistent rhinitis was managed with pharmacotherapy including intranasal steroids and oral antihistamines. Intranasal steroids were kept at the same dose during the study and antihistamines were used as required.
  Arms: Pharmacotherapy

SUMMARY:
While allergen specific immunotherapy (SIT) is highly effective for allergic diseases in children, the underlying immunological mechanisms are unclear. Regulatory T (Treg) cells may be crucial in induction of tolerance.

Our aim was to investigate the role of CD4+CD25+Foxp3+ T cells and IL-10-secreting type I T regulatory (Tr1) cells in the response to one year of cluster SIT to Dermatophagoides pteronyssinus for allergic rhinitis in children.

CD4+CD25+Foxp3+regulatory T cells and IL-10-secreting type I T regulatory (Tr1) cells were analyzed in children allergic to Dermatophagoides pteronyssinus during one year cluster specific immunotherapy (SIT) in a prospective and randomized study. Peripheral blood mononuclear cells (PBMCs) were collected from 25 children receiving SIT and 21 receiving pharmacotherapy. The frequencies of CD4+CD25+Foxp3+ T cells and allergen-specific IL-10+IL-4-, IFN-γ+IL-4-, IL-4+IFN-γ-CD4+ T cells were measured by flow cytometry. Production of IL-4, IFN-r, and IL-10 in supernatants from allergen-stimulated PBMC culture was measured by ELISA. Finally, the suppressive effect of CD4+CD25highTreg cells from both groups was estimated.

DETAILED DESCRIPTION:
Patients The design was a one-year, randomized open-label parallel group study in which patients were randomized in a 1:1 ratio to receive SIT with Dermatophagoides pteronyssinus extract (Alutard SQ, ALK-Abello', Hørsholm, Denmark) or to observe with standard pharmacotherapy (control group).

The study participants included 50 house dust mite (HDM)-allergic children aged 9-13, who received SIT with Dermatophagoides pteronyssinus (Der p) extract for one year. These were compared with 21 HDM-allergic children aged 9-14 who served as controls. All children were of Han nationality and were recruited from the allergy clinic of Beijing TongRen Hospital. They had a history of HDM-induced moderate or severe rhino-conjunctivitis of at least three years duration. Each patient also had a positive skin prick test (SPT) result for Der p (ALK-Abello', Hørsholm, Denmark) with a wheal diameter of at least 6 mm, and were positive for specific immunoglobulin E (IgE) to Der p (Pharmacia CAP System, Pharmacia Diagnostics, Uppsala, Sweden), with a RAST value of at least 0.7 kU/L. Children with a history of asthma or atopic dermatitis were excluded. The children undergoing immunotherapy were matched to atopic donors for age, sex, SPT response to Der p, total IgE and specific IgE to Der p levels (Table 1). The study protocol was approved by our institutional review board for human studies and informed consent was obtained from all subjects.

Immunotherapy protocol Children undergoing subcutaneous immunotherapy were given Dermatophagoides pteronyssinus extract (Alutard SQ, ALK-Abello, Hørsholm, Denmark) according to a cluster protocol which we have described previously[15]. In the first six weeks, children underwent visits for up-dosing, receiving two injections one hour apart with an increasing dose every week. The highest concentration, given in the sixth week, had an allergenic activity of 100,000 SQ/ml and contained 9.8 μg/ml Der p1. After week six, the dosing interval was increased to one month and maintained until the end of the first year. For patients randomized to non-SIT group, persistent rhinitis was managed with pharmacotherapy including intranasal steroids and oral antihistamines. Intranasal steroids were kept at the same dose during the study and antihistamines were used as required. Blood samples were taken at the baseline and after one year treatment in both groups.

Clinical evaluation Symptoms of AR children were assessed by the Total 5 Symptom Score (T5SS), which includes rhinorrhea, sneezing, nasal congestion, and nasal and ocular pruritus. Each symptom was scored on a scale of 0-3 (0 = none, 3 = severe). Medication use was scored and recorded daily, as described previously [16]. Arbitrary scores were attributed to the drugs used (0.75 points for 1 puff of nasal corticosteroids and 1 points for 1 tablet of antihistamine). Patients were instructed to use local steroids only (plus antihistamines if they did not improve symptoms) and to report each administration or variation of the initial drug therapy in the diary. Patients were also instructed to stop drugs at least 7 days before blood sampling.

Flow cytometry Peripheral blood was obtained by venous puncture and collected into preservative-free heparin. Peripheral blood mononuclear cells (PBMCs) were isolated by means of Ficoll-Plaque Plus density gradient centrifugation (Amersham Biosciences, NJ, USA). For intracellular detection of cytokine, PBMCs (2 × 106 cells/mL) were stimulated with 10 μg/mL Der p1 (D. pteronyssinus major allergen 1, Indoor Biotechnologies, United Kingdom) for 24 hours. Twenty-five ng/mL phorbol 12-myristate 13-acetate (PMA), 1 μg/mL ionomycin and 1.7 μg/mL monensine were added at 37 °C for the final four hours of stimulation (all from Sigma, Missouri, USA).

For flow cytometry, PBMCs were surface stained at room temperature for 20 minutes with anti-CD4-PerCP and anti-CD25-PE, or isotype control (mouse IgG1-PerCP or IgG1-PE) (all from Beckman Coulter, CA, USA). For intracellular staining of Foxp3, cells were fixed and permeabilized with Foxp3 fixation/permeabilization buffer, then stained with anti-human Foxp3-FITC or isotype control (IgG1-FITC) (all from BioLegend, CA, USA). For the intracellular cytokine analysis, Der p1-stimulated PBMCs were surface stained with anti-CD3-APC and anti-CD8-PerCP, and fixed with 4% paraformaldehyde/PBS. After being permeabilized using FACS Permeabilizing Solution (BD Pharmingen, CA, USA), cells were incubated for 30 minutes at room temperature with anti-IL-4-PE plus anti-IFN-γ-FITC, or anti-IL-10-PE plus anti-IL-4-FITC, and each antibody was matched with a respective isotype IgG1 as a control (all from BD Pharmingen). Different T subsets were selected for detailed phenotypic analysis as follows: (1) Th1 cells: IFN-γ+IL-4-CD3+CD8- T cells; (2) Th2 cells: IL-4+IFN-γ-CD3+CD8- T cells; and (3) Tr1 cells: IL-10+IL-4-CD3+CD8- T cells. For each analysis, at least 20,000 events were collected. Analysis was conducted using a FACSCalibur flow cytometer (BD Biosciences, NJ, USA).

ELISA PBMCs were resuspended at 2 × 106 cells/mL in RPMI-1640 medium and stimulated with 10 μg/mL Der p1 (D. pteronyssinus major allergen 1, Indoor Biotechnologies, United Kingdom). Cultures were incubated for 6 days at 37 ºC in a humidified incubator containing 5% CO2. Supernatants from allergen-stimulated PBMCs cultures were assayed for the presence of IFN-γ, IL-4, and IL-10 by means of ELISA (R&D Systems, Minneapolis, USA).

Isolation of CD4+CD25high Treg cells Heparinized blood was obtained from each of eight recruited SIT-treated children and eight AR controls for cell isolation and functional analysis. After non-CD4+ cells in the PBMCs were removed by LD column with a biotin-antibody cocktail and antibiotin microbeads, CD4+ T cells were isolated from the PBMCs by negative selection, and CD4+CD25+ T cells were positively selected from the CD4+ T cells. Finally, CD25- fractions were recovered using a MS-magnetic column using a human CD4+CD25+ regulatory T cell isolation kit according to the manufacturer's instructions (Miltenyi Biotec, Germany). Cells with the highest CD25 expression (CD25high) were selected through incubation with a limiting quantity of anti-CD25 antibody beads (2 μl of anti-CD25 beads/107 cells)[17]. The mean purity of the isolated CD4+ was 95% (93-97%) and 76% (72-88%) for CD4+CD25high T cells being Foxp3-positive.

Suppressive capacity of CD4+CD25high Treg cells To evaluate the suppressive capacity of CD4+CD25high Treg cells, cell proliferation and cytokine were analyzed. CD4+CD25- T cells (responders) alone or mixed CD4+CD25- T cells and CD4+CD25high T cells (suppressors) at a ratio of 2:1 were cultured in a final volume of 200 µl RPMI-1640 medium with 10 µg/ml Der p1. Cultures were incubated for 6 days at 37 ºC in a humidified incubator with 5% CO2. Autologous irradiated PBMCs (3000 rad) were added at 2 × 105 as antigen-presenting cells to CD4+CD25- T cell cultures. In all cases, triplicate medium wells were included as negative controls. At day six, 100 µl of supernatant was removed for Th1 and Th2 cytokine (IFN-γ and IL-4) analysis with an ELISA kit (R&D Systems, Minneapolis, USA). Cell proliferation of CD4+CD25- T cells was then assessed using a WST-8 (modified tetrazolium salt) cell proliferation kit (Cell Counting Kit-8, Dojin, Japan) according to the manufacturers' protocols. The proliferation result was expressed as absorbance at 450nm of the culture medium.

Statistics Statistical significance between groups was analyzed using a Mann-Whitney test. The significance of intra-group pre- and post-therapy changes were determined using a nonparametric Wilcoxon matched pairs test. The correlation coefficient r was generated using the Pearson correlation. All analyses were performed using SPSS version 13.0 statistical software. A 5% significance level was used (α = 0.05), power (1- β) equal to 90%. All tests were 2-tailed, and P values of less than 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Allergic rhinitis
* Han nationality
* Had a history of HDM-induced moderate or severe rhino-conjunctivitis of at least three years duration
* Had a positive skin prick test (SPT) result for Der p (ALK-Abello', Hørsholm, Denmark) with a wheal diameter of at least 6 mm
* Were positive for specific immunoglobulin E (IgE) to Der p (Pharmacia CAP System, Pharmacia Diagnostics, Uppsala, Sweden), with a RAST value of at least 0.7 kU/L

Exclusion Criteria:

* Clinical diagnosis of asthma

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Symptom evaluation | Clinical results were based on the patient self-evaluation scores obtained at the beginning and after 3, 6 and 12 months of treatment.
  Symptoms of AR children were assessed by the Total 5 Symptom Score (T5SS), which includes rhinorrhea, sneezing, nasal congestion, and nasal and ocular pruritus. Each symptom was scored on a scale of 0-3 (0 = none, 3 = severe).

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, M.D, Principal Investigator — Beijing Institiute of Otolaryngology
Locations (1):
- the allergy clinic of Beijing TongRen Hospital, Beijing, China